CLINICAL TRIAL: NCT03270137
Title: Cognitive, Behavioral and Functional Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Potential Alzheimer Disease: Two Treatment Modalities Comparison
Brief Title: Repetitive Transcranial Magnetic Stimulation in Patients With Alzheimer Disease
Acronym: AD-EMTr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Ruth Alcala Lozano, Principal Investigator, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIC-16-001
Record Dates: First submitted 2017-08-21; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer Disease; Transcranial Magnetic Stimulation
Keywords: Alzheimer Disease; rTMS; Cognition; Behavioral Symptoms; Functionality
MeSH Terms: conditions — Alzheimer Disease; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Masking Description: Single Blind (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condition A: rTMS on L-DLPFC (Active Comparator): Repetitive transcranial magnetic stimulation- IDLPFC. The intervention will be rTMS delivered on left dorsolateral prefrontal cortex (L-DLPFC).
  Every patient will receive 15 rTMS sessions (in weekdays) along three weeks at 5 Hz of frequency and at its 100% of motor threshold. Each session will consist of 30 trains separated by 10 seconds inter-train interval and 1500 total pulses per session.
  Equipment to rTMS includes a Magpro R30 stimulator (Magventure, Denmark) with an 8-shape coil model MCF-B70.
  Interventions: Device: repetitive transcranial magnetic stimulation- IDLPFC
- Condition B: rTMS on six regions (Active Comparator): Repetitive transcranial magnetic stimulation - Six regions. Two sub-conditions will alternate each session, starting with day 1: rTMS on Broca and Wernicke area and lDLPFC and then day 2: rTMS on left and right parietal association cortex (lPAC; rPAC) and right dorsolateral prefrontal cortex (rDLPFC).
  Patients will receive 15 intervention sessions (in weekdays) along three weeks at 5 Hz frequency and 100% of motor threshold. Each area will receive 10 trains (500 pulses) separated by 10 seconds of inter-train interval that correspond to 1500 total pulses per session.
  Equipment to rTMS includes a Magpro stimulator (Dantec, Denmark) with an 8-shape coil model MC-B70.
  Interventions: Device: repetitive transcranial magnetic stimulation - Six regions

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation- IDLPFC — Repetitive transcranial magnetic stimulation (rTMS) at 5Hz administered over left dorsolateral prefrontal cortex (lDLPFC). Repetitive transcranial magnetic stimulation (rTMS) at 5Hz administered over left dorsolateral prefrontal cortex (lDLPFC) compared to six regions protocol, divided in two sub-conditions: day 1 (Broca area, Wernicke area and lDLPFC) alternated by day 2 (left and right parietal association cortex, and right dorsolateral prefrontal cortex [rDLPFC]). Main outcomes will be evaluated at ending of 15 rTMS sessions and 4 weeks after.
  Arms: Condition A: rTMS on L-DLPFC
Device: repetitive transcranial magnetic stimulation - Six regions — Repetitive transcranial magnetic stimulation (rTMS) at 5Hz administered on six regions protocol, divided in two sub-conditions: day 1 (Broca area, Wernicke area and lDLPFC) alternated by day 2 (left and right parietal association cortex, and right dorsolateral prefrontal cortex [rDLPFC]). Main outcomes will be evaluated at ending of 15 rTMS sessions and 4 weeks after.
  Arms: Condition B: rTMS on six regions

SUMMARY:
Randomized clinical trial, comparative and single blind aims to determine effects on cognition, psychological and behavioral symptoms and functionality of 5 Hz repetitive transcranial magnetic stimulation (rTMS) administered over left dorsolateral prefrontal cortex (lDLPFC) compared to six regions protocol, divided in two sub-conditions: day 1 (Broca area, Wernicke area and lDLPFC) alternated by day 2 (left and right parietal association cortex, and right dorsolateral prefrontal cortex [rDLPFC]). Main outcomes will be evaluated at ending of 15 rTMS sessions and 4 weeks after.

DETAILED DESCRIPTION:
Alzheimer disease (AD) is a neurodegenerative disorder characterized by progressive cognitive decline that affects behavior and daily functionality. Its etiology is unknown and treatment efficacy is partial. Repetitive transcranial magnetic stimulation has been suggested as a potential treatment as of several trials has revealed improvements in language, episodic memory, psychological and behavioral symptoms in dementia as well as functionality using different experimental designs, stimulation parameters and cortical targets comparisons. However, it remains to determine the most effective modality, comparing outcomes with cortical targets poorly studied and how much the effects last. The main objective of this study is to determine which of two stimulation modalities provides a better cognitive and behavioral effect also on functionality in patients with potential diagnosis of AD, administered over lDLPFC (Condition A) and a six areas condition (Condition B) in which are alternated two sub-conditions (Day 1: Broca and Wernicke areas and lDLPFC, and Day 2: bilateral parietal association cortex and rDLPFC) along 15 sessions and 1500 pulses per session.

For this purpose, will be randomized 22 patients with potential diagnosis of AD (according to DSM-5) to both stimulation conditions (11 patients to each condition). The rTMS will be administered at 5 Hz and 1500 pulses per session (30 trains and 10 seconds inter-train interval) along 15 sessions with a post-treatment evaluation at 4 weeks comparing: time response, post-treatment effects and 4 weeks effects.

To evaluate clinical response among stimulation conditions will be used Alzheimer´s Disease Assessment Scale COGNITIVE (ADAS-cog), Cumming's Neuropsychiatric Inventory (NPI), Yesavage Geriatric Depression Scale (GDS), Interview for Deterioration-in-daily Living Activities in Dementia (IDDD) and Clinical Global Impression (CGI). The modified version of Mini Mental State (MMSE-FOLSTEIN) will be applied in the same time points of other evaluations also at the session 5 and 10. Other interest variables are: age, sex, civil status, education, occupation, time and type of pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with file number at National Institute of Psychiatry "Ramón de la Fuente Muñiz".
* Scholarship of at least 5 years or above.
* Dementia diagnosis established by clinical examination made by their responsible physician, according the Diagnose Criteria for Alzheimer Disease for possible, mild or moderate according to DSM-5. Severity will be stratified with Mini-Mental State (MMSE-FOLSTEIN): as a) mild: 21-26 and b) moderated 15-20 points; in addition, with Reisberg Global Deterioration, the states from 2 to 4 that correspond a cognitive deficit mild and moderated.
* In the case of concomitant treatment with memantine or acetylcholinesterase inhibitors, the patient should have taken it for at least 6 months prior to study.
* In the case of other pharmacological treatments for psychiatric conditions, for example, antidepressants, anxiolytic or antipsychotics, the patient should have taken stable doses for at least 2 months.
* Patients with another no-psychiatric comorbidity should be stable (according to diagnostic criteria and supported by laboratory studies or metric assessments).
* Every patient should have a caregiver (for example, spouse, a relative or a professional caregiver) along the study who could stay with the patient at least 10 hours/week.
* Signing of informed consent by patient and caregiver.
* Patients and caregivers who can attend in weekdays, along three weeks assessments and treatment sessions at National Institute of Psychiatry "Ramón de la Fuente Muñiz".

Exclusion Criteria:

* Patients with severe agitation symptoms or difficulties to cooperate with the study.
* Patients with history of epilepsy.
* Patients with sudden onset of apoplexy, focal neurologic findings as hemiparesis, sensory loss, visual field deficit and lack of coordination in the legs in early stages of disease.
* Convulsion or walking disorder at onset or very early stages of the disease.
* Patients with history of severe psychiatric disorders.
* Patients with alterations in a conventional electroencephalogram (paroxysmal phenomena identified by a specialized clinical neurophysiologist).
* Patients with pacemaker or implanted metallic intracranial objects.

Elimination criteria:

* Decision of patient or caregiver to left the study.
* Modification in doses or pharmacological treatment prior to start the study.
* Patients with new clinical findings and who require complementary pharmacological treatment.
* Presence of adverse events that could affect health and could limit maintain the patient in treatment.
* Exacerbation of cognitive or behavioral symptoms during the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes on cognitive functioning (ADAS-cog) | Baseline, Post rTMS treatment: at week 3, and at week 4.
  ADAS-cog is cognitive testing instrument to measure severity. It explores 11 domains including memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD.

SECONDARY OUTCOMES:
Changes on cognitive effects (Mini Mental State) | Baseline, every week for 3 weeks during rTMS treatment and at the 4th week after treatment.
  This instrument gives scores to orientation in time and space, registration information (three words) and recovering, attention, calculation, language (denomination, repetition, understanding of complex orders, reading and writing) and finally visuoconstruction (two overlapping diamonds).
Changes on behavioral symptoms (NPI) | Baseline, Post rTMS treatment: at week 3, and at week 4.
  This is a diagnostic instrument to determine the presence of behavioral symptoms. It measures frequency and severity of symptoms in the last month and the overload for the caregiver. This test divides behavioral symptoms in: delirium, hallucinations, agitation or aggressivity, anxiety, euphoria, apathy, irritability/lability, disinhibition, aberrant motor behavior, sleep and appetite/feeding.
Changes on depression symptoms (GDS-Yesavage) | Baseline, Post rTMS treatment: at week 3, and at week 4.
  Repeated application allows to evaluate changes in the geriatric depression evolution.
Changes on effects on functionality (IDDD) | Baseline, Post rTMS treatment: at week 3, and at week 4.
  This is an instrument designed to evaluate functionality in dementia. It evaluates self-care and complex activities.
Changes on Clinical Global Impression (CGI) | Baseline, Post rTMS treatment: at week 3, and at week 4.
  Standardized and descriptive scale, it gives qualitative information to identify changes in the illness through measuring severity of clinical picture and improvements triggered by treatments (change in the time) as well as treatment efficacy.

IPD SHARING:
Plan to Share IPD: Undecided